CLINICAL TRIAL: NCT07391852
Title: Circadian Light Exposure Adjustment for Restfulness
Acronym: CLEAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00005764: CLEAR; K01HL181331 (NIH)
Record Dates: First submitted 2026-01-07; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Sleep Onset Latency
Keywords: Behavioral sleep problems; Circadian phase; sleep onset latency; Early childhood; dim light melatonin onset (DLMO); Evening light exposure; Light intervention

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are blinded to study condition. Research staff are aware of assignment after baseline assessments. Laboratory technicians conducting melatonin assays are blinded to study hypotheses and participant condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Amber Tinted Glasses (Experimental): Wearing "blue-blocker" glasses (lenses that filter out the blue portion of the visible spectrum) can reduce the melatonin suppression and alertness effects of evening light exposure in both adults and adolescents, as well as advance the timing of the circadian clock and sleep onset, compared with participants wearing placebo lenses. This intervention will examine their efficacy in advancing young children's sleep and circadian timing. Children will be given a pair of glasses (Block Blue Light), with amber-tinted lenses (advertised as blocking 100% of light from 380-550 nm. Children will wear the glasses starting 1 h before parent's selected bedtime each evening across the two-week intervention. Parents will also complete a daily diary detailing when the glasses are worn.
  Interventions: Device: Amber Tinted Glasses
- Clear Glasses (Sham Comparator): The sham comparator consists of the same protocols for the amber-tinted glasses, except that children will wear a pair of glasses with clear lenses (advertised as blocking 50% of light from 400-500 nm), which are significantly less effective at blocking short-wavelength light.
  Interventions: Device: Clear Glasses
- Smart Lightbulbs (Experimental): The presence of more blue light in the home is associated with later circadian timing in both school-aged children and adults. This intervention will adjust the evening home lighting environment to be less stimulating to children's circadian clocks. Smart light bulbs (dimmable and color tunable LED bulbs) will be installed in participants' homes light fixtures, or in the child's bedroom, bathroom, as well as areas the child is likely to spend time in after dinner (i.e., living room, playroom). The researchers will program the lights to transition to a lower CCT and dimmer intensity to achieve the recommended evening mEDI of 10 lux starting 1 h before the child's parent-selected bedtime.
  Interventions: Device: Smart Lightbulbs

INTERVENTIONS:
Device: Amber Tinted Glasses — Children will wear amber-tinted glasses in the evening hours before bedtime to reduce exposure to short-wavelength (blue) light. The glasses are intended to reduce circadian disruption associated with evening light exposure.
  Arms: Amber Tinted Glasses
Device: Clear Glasses — Children will wear clear glasses in the evening hours before bedtime. This sham intervention controls for wearing glasses without reducing light exposure.
  Arms: Clear Glasses
Device: Smart Lightbulbs — Smart light bulbs will be installed in the child's home and programmed to reduce short-wavelength light exposure during evening hours before bedtime.
  Arms: Smart Lightbulbs

SUMMARY:
Many young children are exposed to light int he evening hours before bedtime. Children's biological clocks are highly sensitive to evening light exposure, which can delay the timing of the clock and make it harder to fall asleep. The purpose of this study is to test three strategies (adjustment to home lighting, amber-tinted glasses, clear glasses) to reduce evening light exposure in children ages 5-6 years with parent-reported sleep onset difficulties in order to improve their sleep and the timing of their biological clock. This study takes place over approximately 5 weeks. After baseline assessments of children's sleep timing, light exposure, cognition, and circadian rhythms, they will be randomly assigned to one of three interventions to reduce evening light exposure for two weeks. After the two-week intervention period, the baseline measures are repeated and parents are interviewed about their and their child's experiences with the intervention.

DETAILED DESCRIPTION:
Evening sleep difficulties are common in young children and can contribute to behavioral and health problems. Sleep timing is regulated in part by the circadian clock, which is highly sensitive to light exposure. Light in the hour before bedtime can suppress melatonin, delay circadian timing, and make it harder for children to fall asleep. Despite evidence of high circadian sensitivity to evening light, few studies have tested interventions to improve sleep timing in early childhood using light-based strategies.

This study evaluates the feasibility, acceptability, and preliminary efficacy of two light-mitigation strategies to advance sleep and circadian timing in children aged 5 to 6 years with parent-reported sleep onset difficulties. Children will participate in a five-week study consisting of baseline assessments, a two-week intervention period, and post-intervention assessments. Parents of enrolled children will provide written informed consent for their child's participation. Children are under age 7 years and are not required to provide formal assent.

Baseline assessments will include sleep timing, duration, and quality measured via actigraphy, circadian phase assessed with salivary dim-light melatonin onset (DLMO), parent-reported sleep behaviors, and a cognitive battery. Children will then be randomly assigned to one of three interventions: (1) smart home lighting to reduce evening short-wavelength light, (2) amber-tinted glasses worn in the hour before bedtime, or (3) clear glasses as a sham control. Interventions will last two weeks, with adherence monitored throughout.

After the intervention, all assessments will be repeated, and parents will participate in structured interviews to report on the feasibility and acceptability of the assigned strategy. Exploratory measures will include baseline pupillary light response to examine individual differences in photosensitivity as potential moderators of intervention effects.

Data from this study will inform the feasibility and acceptability of light-based interventions in young children (Aim 1), provide preliminary evidence of effects on sleep and circadian timing (Aim 2), and explore whether photosensitivity moderates response to the interventions (Exploratory Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion requires that children are aged 5.0-6.9 years at the time of enrollment with a parent-reported sleep onset of ≥ 60 min after parents' desired bedtime at least three nights per week.

One adult parent of each participating child will also take part in the study. Parents must be able to provide consent for themselves and their child and to complete the interview at the end of the study.

Exclusion Criteria:

* Children are excluded for the following reasons:

  * All sleep disorders as indicated on the telephone screener or by clinical cut-off scores on the Children's Sleep Habits Questionnaire (CSHQ), except for insomnia or DSWPD as features of these disorders are directly targeted by the intervention. Secondary analyses will explore if outcomes differ among participants with or without parent-reported symptoms consistent with these diagnoses.
  * Physical abilities that interfere with assessments (e.g., visual impairment), developmental disabilities (e.g., autism, attention-deficit/hyperactivity disorder (ADHD), pervasive developmental disorder), epilepsy or other neurological disorders, metabolic disorders, medical conditions that commonly require treatments or assessments during the night (e.g., cancer, diabetes, active asthma), current infection or lead poisoning; a head injury involving loss of consciousness in the past 6 months.
  * Current use of medications affecting daytime sleepiness, the circadian system, or light sensitivity.
  * Eye disorders or color blindness (determined with Ishihara Color Vision Test); corrected vision with eyeglasses is permitted.

Ages: 60 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility | Throughout the two-week intervention period.
  Feasibility will be assessed using adherence/compliance rates to assigned intervention protocols.
Acceptability | Week 5
  Acceptability will be assessed using parent-reported qualitative interviews conducted post-intervention.

SECONDARY OUTCOMES:
Circadian Timing | Assessed once in Week 2 and once in Week 5
  Dim light melatonin onset, a measure of circadian timing, will be assessed via saliva samples.
Sleep Timing | Throughout the 5 week protocol
  Throughout the duration of the study, the child will wear a wrist actigraph which records sleep timing and light exposure. The actigraph is a watch-size monitor worn on the non-dominant wrist, providing continuous imputation of sleep-wake states via arm activity. These data will be used to examine changes in habitual sleep timing, sleep onset latency.
Light Exposure | Throughout the 5 week protocol.
  Measured by the wrist-worn actigraph watch in 1-min epochs throughout data collection. These data provide an objective measure of the child's light exposure throughout the protocol (including compliance with the home lighting intervention) and will be used to examine changes in habitual light exposure.
Sleep-Related Behaviors | Assessed once in Week 1 and once in Week 5
  Change in parent-reported sleep behaviors assessed via validated questionnaires.

OTHER OUTCOMES:
Pupillary Light Response | Baseline
  Baseline pupillary light response will be assessed as a measure of individual differences in photosensitivity.
Cognitive Functioning | Assessed once in Week 1 and once in Week 5
  Change in cognitive performance from pre- to post-intervention assessed using a standardized cognitive battery (NIH Toolbox).

CONTACTS AND LOCATIONS:
Overall Officials: Lauren E Hartstein, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
No identifiable data will be shared. Only de-identified study data will be made available for research purposes.

REFERENCES:
- [Background] Werner H, Lebourgeois MK, Geiger A, Jenni OG. Assessment of chronotype in four- to eleven-year-old children: reliability and validity of the Children's Chronotype Questionnaire (CCTQ). Chronobiol Int. 2009 Jul;26(5):992-1014. doi: 10.1080/07420520903044505. PMID 19637055
- [Background] LeBourgeois MK, Harsh JR. Development and psychometric evaluation of the Children's Sleep-Wake Scale<sup/> Sleep Health. 2016 Sep;2(3):198-204. doi: 10.1016/j.sleh.2016.04.001. PMID 28066802
- [Background] Zerbini G, Kantermann T, Merrow M. Strategies to decrease social jetlag: Reducing evening blue light advances sleep and melatonin. Eur J Neurosci. 2020 Jun;51(12):2355-2366. doi: 10.1111/ejn.14293. Epub 2018 Dec 13. PMID 30506899
- [Background] van der Lely S, Frey S, Garbazza C, Wirz-Justice A, Jenni OG, Steiner R, Wolf S, Cajochen C, Bromundt V, Schmidt C. Blue blocker glasses as a countermeasure for alerting effects of evening light-emitting diode screen exposure in male teenagers. J Adolesc Health. 2015 Jan;56(1):113-9. doi: 10.1016/j.jadohealth.2014.08.002. Epub 2014 Oct 3. PMID 25287985
- [Background] Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000 Dec 15;23(8):1043-51. PMID 11145319
- [Background] Lebourgeois MK, Wright KP Jr, Lebourgeois HB, Jenni OG. Dissonance Between Parent-Selected Bedtimes and Young Children's Circadian Physiology Influences Nighttime Settling Difficulties. Mind Brain Educ. 2013 Dec;7(4):234-242. doi: 10.1111/mbe.12032. PMID 24535929
- [Background] Hartstein LE, Wong SD, Abbas L, Choubai S, Wilson JN, Jablin T, LeBourgeois MK. Creating the Cave: Conducting Circadian Science in Early Childhood. Clocks Sleep. 2023 Feb 20;5(1):85-93. doi: 10.3390/clockssleep5010009. PMID 36810846
- [Background] Hartstein LE, Diniz Behn C, Wright KP Jr, Akacem LD, Stowe SR, LeBourgeois MK. Evening Light Intensity and Phase Delay of the Circadian Clock in Early Childhood. J Biol Rhythms. 2023 Feb;38(1):77-86. doi: 10.1177/07487304221134330. Epub 2022 Nov 22. PMID 36415902
- [Background] Hartstein LE, Behn CD, Akacem LD, Stack N, Wright KP Jr, LeBourgeois MK. High sensitivity of melatonin suppression response to evening light in preschool-aged children. J Pineal Res. 2022 Mar;72(2):e12780. doi: 10.1111/jpi.12780. Epub 2022 Jan 8. PMID 34997782

DOCUMENTS (2):
  • Study Protocol (2025-12-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT07391852/Prot_000.pdf
  • Informed Consent Form (2025-12-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT07391852/ICF_001.pdf